CLINICAL TRIAL: NCT05706961
Title: Effect Of Power Walking On Quality Of Life In Post CABG Patient Undergoing Phase 2 Cardiac Rehabilitation
Brief Title: Power Walking On Quality Of Life In Post CABG Patient Undergoing Phase 2 Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/01374 Awais Ahmed
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power Walking (Experimental)
  Interventions: Other: Power Walking
- Standardized Outpatient Cardiac Rehabilitation (Active Comparator)
  Interventions: Other: Standardized Outpatient Cardiac Rehabilitation

INTERVENTIONS:
Other: Power Walking — For 1- 2 Week 60% of the target heart rate with 5,000 to 7,500 steps/day Total 30 min Session The exercise intensity was set at 60% of the target heart rate during the first 2 weeks.
  For 3- 4 week 70 % of the target heart rate with 7,500 to 10,000 steps/day Total 30 min Session B) Progressive increase walk according to 6MWD as improved Low intensity
  Arms: Power Walking
Other: Standardized Outpatient Cardiac Rehabilitation — For 1- 2 week Standardized Outpatient Cardiac Rehabilitation (includes warm up of 5 min, aerobic 60 % of of target heart rate, resistive ex with 1- 3 kg of weight for 20 min and 10 min of cool down)
  For 3 - 4 week Standardized Outpatient Cardiac Rehabilitation (includes warm up of 5 min, aerobic 70 % of target heart rate, resistive ex with 2- 3 kg of weight for 20 min and 10 min of cool down)
  Arms: Standardized Outpatient Cardiac Rehabilitation

SUMMARY:
To determine the effect of power walking on quality of life in Post CABG population undergoing phase 2 cardiac rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subject
* Age will be from 50 to 70
* Four weeks after CABG surgery patient are eligible to participate
* Patient able to walk on Treadmill with Cardiac symptoms stable or absent
* Appropriate HR response to exercise

Exclusion Criteria:

* Those patients with contraindications to exercise or clinical risk factors, such as musculoskeletal, neurological, pulmonary or metabolic disorder were all excluded from the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Heart Quality of Life questionnaire | 4th weeks
  Changes from baseline to 4 week, The 14 items in the HeartQoL scale form a bi-dimensional questionnaire with a 10-item HeartQoL physical subscale and a 4-item HeartQoL emotional subscale that provides a global assessment and evaluation of how much a patient with angina, MI, or heart fail.

SECONDARY OUTCOMES:
Six Minute Walk Test (6MWT) | 4th week
  Changes from baseline to 4 week, The 6MWT can be used in preschool children (2-5 years), children (6-12 years) adults (18-64 years), elderly adults (65+) with a wide range of diagnoses including. The test was initially designed to help in the assessment of patient with cardiopulmonary is
BORG Rating of Perceived exertion | 4th Week
  Changes from baseline to 4 week, The Borg RPE Scale is a 15-point scale (6 to 20) used to rate subjective experiences during physical exertion. This subjective load scale can help estimate load symptoms, such as the degree of exertion, the degree of load and fatigue. The Borg scale among
Pulse rate | 4th Week
  Changes from baseline to 4 week, Pulse rate will be measured through the Pulse Oximeter in beats per min before and after the exercise for the patient safety during exercise
Liebowitz Social Anxiety Scale | 4th Week
  Changes from baseline to 4 week, The LSAS is a 24-item scale that assesses fear of social situations and avoidance throughout the previous week. It includes 11 things that deal with social contact and 13 ones that deal with public performance. A physician rates each item on two 4-point L

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Women Institute of Rehabilitation Sciences (WIRS) and Jinnah International Hospital, Abbottābād, Khyber PkahtoonKhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No